CLINICAL TRIAL: NCT04060797
Title: Endovascular Denervation Improves Limb Ischemia in Patients With Peripheral Artery Disease (ED-PAD)
Brief Title: Endovascular Denervation Improves Limb Ischemia in Patients With Peripheral Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Clinical Professor, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ED-PAD
Record Dates: First submitted 2019-08-16; First posted 2019-08-19 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: PAD

STUDY DESIGN:
Intervention Model Description: Patients were randomly divided into two groups: the endovascular revascularization (ER) group and the ER + endovascular denervation (EDN) group treating with EDN at the site of the distal iliac artery or the proximal superficial femoral artery before ER
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (Other): Treating with balloon dilation or stent implantation only,
  Interventions: Device: PTA
- The EDN group (Experimental): Treating with (Endovascular Denervation) EDN at the site of the iliac artery distal to the superficial femoral artery proximal before balloon dilation or stent implantation.
  Interventions: Device: endovascular denervation; Device: PTA

INTERVENTIONS:
Device: endovascular denervation — Treating with endovascular denervation (EDN) at the site of the iliac artery distal to the superficial femoral artery proximal before balloon dilation or stent implantation
  Arms: The EDN group
Device: PTA — Treating with balloon dilation or stent implantation which were Percutaneous transluminal angioplasty (PTA)

SUMMARY:
Sympathetic overactivity partly promotes the development of peripheral artery disease which mainly leads to ischemia of the lower limbs. Endovascular arterial denervation (ED) is a minimally invasive technique which could deliver Radiofrequency energy by a multi-electrode catheter to the Lower limb artery to restore Sympathetic activity. The purpose of this study is to evaluate the effects of multi-electrode radiofrequency ablation system on lower limb ischemia with PAD.

DETAILED DESCRIPTION:
Peripheral arterial disease(PAD) show insufficient blood supply of diseased limbs, which causes intermittent claudication of lower limbs, reduced skin temperature, pain, and chronic progressive disease that still produces ulcer or necrosis. Some clinical studies have shown Sympathetic overactivity in the lower arterial ischemic disease. The multi-electrode radiofrequency ablation system can significantly reduce the excitability of sympathetic nerve, restore the normal response of sympathetic nerve, relieve the pain and discomfort of patients, effectively improve the symptoms of lower limb ischemia, and improve the quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

1. eligible subjects aged 18-75 years,
2. clinically confirmed PAD in the lower extremities,
3. Rutherford category II-VI.

Exclusion Criteria:

1. thrombolytic therapy performed within 30 days,
2. patients who had undergone vascular bypass surgery before this study,
3. allergy or contraindication of antiplatelet drugs, anticoagulants, thrombolytic drugs and contrast agents,
4. patients with obvious bleeding tendency, coagulation dysfunction, hypercoagulability and blood system diseases,
5. serious liver and kidney diseases,
6. history of hemorrhagic stroke within last month or ischemic stroke or transient ischemic attack within 2 weeks,
7. pacemaker implants,
8. patients who are pregnant, breast-feeding or planning pregnancy,
9. expected survival < 24 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | The Control Group | The EDN Group
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | The Control Group | The EDN Group | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 11
  >=65 years | 12 | 15 | 27
Age, Continuous [Median (Standard Deviation); unit: years] | 67.53 (5.55) | 68.95 (6.76) | 68.24 (6.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 17 | 16 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 19 | 19 | 38
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 19 | 19 | 38
Weight [Median (Standard Deviation); unit: Kg] | 67.95 (9.59) | 68.37 (5.34) | 68.15 (7.76)

OUTCOME MEASURES:

1. Primary Outcome: Change of Ankle Brachial Index (ABI) at 6-month Post-procedure.
Description: The change value was using the ankle brachial index (ABI) at 6-month post-procedure minus the baseline ABI in two group. (the group which have higher change value mean the better result).
  "Ankle Brachial Index (ABI) is the ratio of the blood pressure in the lower legs to the blood pressure in the arms. The normal range for the ankle-brachial index is between 0.90 and 1.30. An index of 0.41 to 0.90 indicates mild to moderate arterial disease and an index of 0.40 and lower indicates severe disease.
Time Frame: From baseline to 6 months post procedure
Measure: Median (Standard Deviation); unit: ratio
Arm/Group | The Control Group | The EDN Group
Number analyzed (Participants) | 19 | 19
ratio | 0.24 (0.15) | 0.44 (0.30)

2. Secondary Outcome: Change of Ankle Brachial Index (ABI) at 3-month Post-procedure.
Description: The change value was using the ankle brachial index (ABI) at 3-month post-procedure minus the baseline ABI in two group. (the group which have higher change value mean the better result) "Ankle Brachial Index (ABI) is the ratio of the blood pressure in the lower legs to the blood pressure in the arms. The normal range for the ankle-brachial index is between 0.90 and 1.30. An index of 0.41 to 0.90 indicates mild to moderate arterial disease and an index of 0.40 and lower indicates severe disease.
Time Frame: From baseline to 3 months post procedure
Measure: Median (Standard Deviation); unit: ratio
Arm/Group | The Control Group | The EDN Group
Number analyzed (Participants) | 19 | 19
ratio | 0.28 (0.19) | 0.48 (0.31)

3. Secondary Outcome: Change of Ankle Brachial Index (ABI) at 1-week Post-procedure.
Description: The change value was using the ankle brachial index (ABI) at 1-week post-procedure minus the baseline ABI in two group. (the group which have higher change value mean the better result) "Ankle Brachial Index (ABI) is the ratio of the blood pressure in the lower legs to the blood pressure in the arms. The normal range for the ankle-brachial index is between 0.90 and 1.30. An index of 0.41 to 0.90 indicates mild to moderate arterial disease and an index of 0.40 and lower indicates severe disease.
Time Frame: From baseline to 1 week post procedure
Measure: Median (Standard Deviation); unit: ratio
Arm/Group | The Control Group | The EDN Group
Number analyzed (Participants) | 19 | 19
ratio | 0.21 (0.20) | 0.28 (0.33)

4. Secondary Outcome: Change of Transcutaneous Oxygen Pressure (TcPO2)
Description: Use the Transcutaneous oxygen pressure (TcPO2) at 6-month post-procedure minus the baseline TcPO2.(the higher the value, the better the results)
Time Frame: From baseline to 6 months post procedure
Measure: Median (Standard Deviation); unit: mmHg
Arm/Group | The Control Group | The EDN Group
Number analyzed (Participants) | 19 | 19
mmHg | 4.95 (13.43) | 15.68 (16.72)

5. Secondary Outcome: Change of Transcutaneous Oxygen Pressure (TcPO2)
Description: Use the Transcutaneous oxygen pressure (TcPO2) at 3-month post-procedure minus the baseline TcPO2.(the higher the value, the better the results)
Time Frame: From baseline to 3 months post procedure
Measure: Median (Standard Deviation); unit: mmHg
Arm/Group | The Control Group | The EDN Group
Number analyzed (Participants) | 19 | 19
mmHg | 5.58 (15.67) | 15.68 (15.82)

6. Secondary Outcome: Change of Transcutaneous Oxygen Pressure (TcPO2)
Description: Use the Transcutaneous oxygen pressure (TcPO2) at 1 week post-procedure minus the baseline TcPO2.(the higher the value, the better the results)
Time Frame: From baseline to 1 week post procedure
Measure: Median (Standard Deviation); unit: mmHg
Arm/Group | The Control Group | The EDN Group
Number analyzed (Participants) | 19 | 19
mmHg | 5.16 (16.93) | 7.12 (15.90)

7. Secondary Outcome: Rutherford Category
Description: Number of Subjects with a decrease in Rutherford Category in 6 months (Rutherford category includes a total of 0-6 grades, grade 0 was asymptomatic, grade 1 was mild intermittent claudication, grade 2 was moderate intermittent claudication, grade 3 was severe intermittent claudication, grade 4 was resting pain, grade 5 was minor tissue defect, grade 6 was tissue ulcer, gangrene. The lower the grade, the better the results)
Time Frame: At 6 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | The Control Group | The EDN Group
Number analyzed (Participants) | 19 | 19
Participants | 17 | 19

8. Secondary Outcome: Rutherford Category
Description: Number of Subjects with a decrease in Rutherford Category in 3 months (Rutherford category includes a total of 0-6 grades, grade 0 was asymptomatic, grade 1 was mild intermittent claudication, grade 2 was moderate intermittent claudication, grade 3 was severe intermittent claudication, grade 4 was resting pain, grade 5 was minor tissue defect, grade 6 was tissue ulcer, gangrene. The lower the grade, the better the results)
Time Frame: At 3 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | The Control Group | The EDN Group
Number analyzed (Participants) | 19 | 19
Participants | 13 | 19

9. Secondary Outcome: Rutherford Category
Description: Number of Subjects with a decrease in Rutherford Category in 1 week (Rutherford category includes a total of 0-6 grades, grade 0 was asymptomatic, grade 1 was mild intermittent claudication, grade 2 was moderate intermittent claudication, grade 3 was severe intermittent claudication, grade 4 was resting pain, grade 5 was minor tissue defect, grade 6 was tissue ulcer, gangrene. The lower the grade, the better the results)
Time Frame: At 1 week post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | The Control Group | The EDN Group
Number analyzed (Participants) | 19 | 19
Participants | 8 | 11

10. Secondary Outcome: NRS Score
Description: Median of numeric rating scale (NRS) scores in 6 months (NRS scores includes a total of 0-10 grades, No pain (0), Mild pain (1 ~ 3), Moderate pain (4 ~ 6), Severe pain (7 ~ 10), the lower the grade, the better the results)
Time Frame: At 6 months post procedure
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | The Control Group | The EDN Group
Number analyzed (Participants) | 19 | 19
score on a scale | 0 [0 to 0] | 0 [0 to 0]

11. Secondary Outcome: NRS Score
Description: Median of numeric rating scale (NRS) scores in 3 months (NRS scores includes a total of 0-10 grades, No pain (0), Mild pain (1 ~ 3), Moderate pain (4 ~ 6), Severe pain (7 ~ 10), the lower the grade, the better the results)
Time Frame: At 3 months post procedure
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | The Control Group | The EDN Group
Number analyzed (Participants) | 19 | 19
score on a scale | 0 [0 to 0] | 0 [0 to 0]

12. Secondary Outcome: NRS Score
Description: Median of numeric rating scale (NRS) scores in 1 week (NRS scores includes a total of 0-10 grades, No pain (0), Mild pain (1 ~ 3), Moderate pain (4 ~ 6), Severe pain (7 ~ 10), the lower the grade, the better the results)
Time Frame: At 1 week post procedure
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | The Control Group | The EDN Group
Number analyzed (Participants) | 19 | 19
score on a scale | 1 [0 to 3] | 0 [0 to 2]

13. Secondary Outcome: Number of Participants With MACE (Major Adverse Cardiovascular Events) and MALE (Major Adverse Limb Events)
Description: MACE (Major adverse cardiovascular events, defined as cerebrovascular accident, myocardial infarction, or death.) and MALE (Major adverse limb events, defined as untreated loss of patency of the revascularization, reintervention on the revascularized segment, or major amputation of the revascularized limb) occurred cases from baseline to 6 months.
Time Frame: From baseline to 6 months
Measure: Number; unit: participants
Arm/Group | The Control Group | The EDN Group
Number analyzed (Participants) | 19 | 19
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline to 6 months
Arm/Group | The Control Group | The EDN Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 1/19 | 2/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The Control Group (N=19) | The EDN Group (N=19)
hematoma at puncture site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
local arterial vasospasm (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT04060797/Prot_SAP_000.pdf